CLINICAL TRIAL: NCT02749240
Title: A Feasibility (Pilot) Study of an Innovative Non-pharmacological Intervention Program in at Risk Youth
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 107708
Record Dates: First submitted 2016-03-22; First posted 2016-04-22 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: At Risk Youth
MeSH Terms: interventions — YES1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Youth Empowerment Seminar, YES! (Other): An 8-week innovative bio-psycho-social program (Youth Empowerment Seminar, YES!) will be offered to at risk youth participating in programs or resources offered by Youth Opportunities Unlimited. The YES! program will be taught in two phases: (1) an active learning phase which consists of four consecutive days (3 hrs/day) of SEL skills taught in a multi-modality interactive format as well as SKY training, and (2) a reinforcement phase which involves weekly follow up sessions (75-90 mins each) for the 7 weeks following the active phase. Two certified instructors from the Art of Living Foundation (Spencer Delisle and Mark Frye) will deliver this training under supervision of Ronnie Newman (RN). After the initial 4 day training, participants will be asked to practice SKY daily for 20-25 minutes in addition to attending the weekly follow up sessions.
  Interventions: Other: Youth Empowerment Seminar, YES!

INTERVENTIONS:
Other: Youth Empowerment Seminar, YES! — An 8-week innovative bio-psycho-social program.

SUMMARY:
At risk youth face various adversities including homelessness, social isolation, substance abuse and other mental illnesses. Thus far, the investigators have successfully partnered on programs of housing, social and recreational interventions in this population. The investigators now wish to assess the feasibility of delivery of an innovative bio-psycho-social intervention, Youth Empowerment Seminar (YES!), developed by their partner, the not-for-profit Art of Living Foundation. Therefore, the aim of this research is to conduct a proof of concept study to determine the feasibility of a novel YES! program as an intervention for at risk youth.

DETAILED DESCRIPTION:
STUDY DESIGN: The proposed is an open-label study with a mixed methods design. Research participants will be thirty youth between the ages of 16-25 years who are currently accessing any resource offered by Youth Opportunities Unlimited, London, ON. Youth will be enrolled in a rolling 8-week YES! Program repeated when adequate group size is achieved (>6 participants). Quantitative and qualitative data will be collected, which will allow for a detailed analysis of the feasibility of YES! as an intervention for youth at risk of homelessness.

STUDY RECRUITMENT: Participants for this study will be recruited through the Youth Action Centre (YAC) of Youth Opportunity Unlimited (YOU), London. Participants will be between 16 and 25 years of age. As this is a pilot study, the investigators have set the sample size to n=30, which is in accordance with current standards for pilot studies. The investigators anticipate to recruit participants at a rate of at least 1 youth/week. Advertisements about the study will be placed throughout YAC (located in the YOU Cornerstone Building, 332 Richmond St., London, ON, N6A 3C3) and Theresa McLachlan, a staff member with YOU Transition Services will provide interested youth with additional information as required. There is no obligation for the youth to take part in the study; all participation is voluntary.

SCREENING AND INITIAL ASSESSMENTS: Potential participants will be screened as per inclusion and exclusion criteria by trained research staff. Immediately prior to the start of the intervention trained raters will meet with participants to obtain demographic information and complete baseline measures of social inclusion, substance use and mental health. Specifically, the following scales will be administered:

1. demographic, service and housing history
2. community integration questionnaire
3. Global Appraisal of Individual Needs- Substance Problem Scale (GAIN-SPS), (GAIN-SPS is a subscale of a biopsychosocial battery that has been designed for clinical and program evaluation and has been validated for use in individuals 11 years of age and older), and
4. Colorado Symptom Index.

ELIGIBILITY:
Inclusion Criteria:

* Between 16-25 years of age
* Currently precariously housed and accessing resources offered by Youth Opportunities Unlimited
* Have sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 30 minutes
* Willing and able to attend 4 initial YES! training sessions and at least 5 of weekly follow up sessions.
* Willing to dedicate 20 minutes/daily to SKY practice

Exclusion Criteria:

* Currently participating in other similar studies
* Currently practicing any type of formal meditation, mindfulness or breathing techniques regularly.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Number of potential participants approached per month. | Through study completion, an average of one year
  The number of potential participants approached per month will be assessed at the end of each month. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Number (proportion) of participants who are successfully screened. | Through study completion, an average of one year
  The number (proportion) of participants who are successfully screened will be calculated at the end of the study. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Number (proportion) of successfully screened participants who enroll. | Through study completion, an average of one year
  The number (proportion) of successfully screened participants who enroll in the study will be calculated at the end of the study. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Rate of participant retention. | Through study completion, an average of one year
  The rate of participant retention will be assessed at the end of the study. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Rate of adherence to study protocol. | Through study completion, an average of one year
  At the end of the study any deviations from the protocol will be examined to determine the rate of adherence to the study protocol. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Proportion of planned ratings that are completed. | Through study completion, an average of one year
  The proportion of completed planned ratings will be calculated at the end of the study. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Intervention cost per case | Through study completion, an average of one year
  The cost per participant of attending the YES! program will be calculated. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Completeness of final data for analysis. | Through study completion, an average of one year
  Study data used for analysis will be examined at the end of the study to assess the completeness of the data. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Length of time to collect all data. | Through study completion, an average of one year
  The length of time to collect all study data will be calculated at the end of the study. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Quality of all collected data. | Through study completion, an average of one year
  At the end of the study the quality of all collected data will be assessed. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Determining if YOU is willing to conduct the study as per study protocol. | Through study completion, an average of one year
  At the end of the study any deviations YOU has made from study protocol will be assessed. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.
Assess if it is safe to apply the intervention. | Through study completion, an average of one year
  At the end of the study all recorded adverse events will be assessed. This information will be used to determine the feasibility of a larger Randomized Controlled Trial (RCT) that would examine the YES! program in at risk youth.

SECONDARY OUTCOMES:
Community integration questionnaire | Change from baseline to Week 4 and 8.
  The Community Integration Questionnaire will be used to assess the social role and community interaction participants have at baseline compared to week 4 and week 8.
Global Appraisal of Individual Needs- Substance Problem Scale (GAIN-SPS) | Change from baseline to Week 4 and 8.
  The Global Appraisal of Individual Needs - Substance Problem Scale (GAIN-SPS) will be used to assess any change in substance problems from baseline to week 4 and week 8.
Colorado Symptom Index | Change from baseline to Week 4 and 8.
  The Colorado Symptom Index will be used to assess any change is psychiatric symptoms from baseline to week 4 and week 8.
demographic, service and housing history (DSSH) | Baseline
  At baseline information will be collected on participants demographics and their service and housing history.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasudev A, Ionson E, Sathiaselan J, Thatipalli A, Chauhan A, Hassan C, Sukhera J, Speechley M, Forchuk C. A feasibility (pilot) mixed methods study of an innovative non-pharmacological breath-based yoga and social-emotional intervention program in an at-risk youth sample in London, Canada. Pilot Feasibility Stud. 2024 Feb 7;10(1):26. doi: 10.1186/s40814-024-01452-0. PMID 38321567